CLINICAL TRIAL: NCT05874466
Title: SenseToKnow STAR Study: A Study of Technologies for Assessing Children's Development
Brief Title: SenseToKnow Autism Screening Device Validation Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00111371; 2P50HD093074 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-05-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Diagnosis; Digital device
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients, 16-37 months of age, recruited through pediatric medical clinics: Consecutive pediatric participants will be recruited and enrolled via > 6 participating sites comprised of pediatric medical clinics (e.g., primary care and family medicine clinics) that are part of the broader Duke University Health System (DUHS) located in North Carolina. Enrollment will proceed until the targets of N = 150 participants diagnosed with autism spectrum disorder and N = 200 without autism are reached.

SUMMARY:
This is a pivotal, prospective, double-blind, study to evaluate the sensitivity and specificity of the SenseToKnow app for the detection of autism spectrum disorder in children 16-36 months of age.

DETAILED DESCRIPTION:
This is a pivotal, prospective, double-blind, study to evaluate the sensitivity and specificity of the SenseToKnow app for the classification of autism spectrum disorder when administered by parents in a sample of patients 16-36 months of age. The trial design is a non-interventional cross-sectional study comparing the SenseToKnow app classification of autism spectrum disorder ("autism") versus non-autism with the patient's diagnostic status based on expert clinical diagnosis in a population of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Duke Health pediatric patient at enrollment
2. 16-<37 months of age at enrollment
3. Parent/legal guardian speaks English or Spanish
4. Parent/legal guardian understands and voluntarily provides informed consent

Exclusion Criteria:

1. Severe motor impairment that precludes study measure completion
2. Known genetic disorders
3. Severe hearing or visual impairment as determined on physical examination according to parent report
4. Acute illnesses likely to prevent successful or valid data collection
5. Uncontrolled epilepsy or seizure disorder
6. History or presence of a clinically significant medical disease, or a mental state that could confound the study or be detrimental to the subject as determined by the investigator
7. Acute exacerbations of chronic illnesses likely to prevent successful or valid data collection
8. Receiving therapies that affect vision
9. Parent/legal guardian and/or investigator believes that the child will be unable/unwilling to sit in the parent's lap to watch the app videos
10. Parent/legal guardian indicates that they or their child is unwilling or unable to complete the app administration, surveys, or diagnostic assessment
11. Participants who are otherwise judged as unable to comply with the protocol by the investigator
12. Any other factor that the investigator feels would make the study measures invalid

Ages: 16 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be patients 16-36 months of age recruited from > 6 sites comprised of pediatric medical clinics that are part of the broader Duke University Health System in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of SenseToKnow for autism detection | Will be calculated based on data from Baseline/Timepoint 1
  Sensitivity = #participants positive for autism on both SenseToKnow and expert clinical diagnosis / #participants positive for autism on both SenseToKnow and expert clinical diagnosis + #participants negative for autism on SenseToKnow who were positive for autism by expert clinical diagnosis
Specificity of SenseToKnow for autism detection | Will be calculated based on data from Baseline/Timepoint 1
  Specificity = #participants negative for autism on both SenseToKnow and expert clinical diagnosis / #participants negative for autism on both SenseToKnow and expert clinical diagnosis + #participants positive for autism on SenseToKnow who were negative for autism by expert clinical diagnosis

SECONDARY OUTCOMES:
Positive Predictive Value of SenseToKnow (with and without adjustment for population prevalence) | Will be calculated based on data from Baseline/Timepoint 1
  The likelihood that a participant with a positive test result has a diagnosis of autism.
Negative Predictive Value of SenseToKnow (with and without adjustment for population prevalence) | Will be calculated based on data from Baseline/Timepoint 1
  The likelihood that a participant with a negative test result does not have a diagnosis of autism
Receiver Operating Characteristic Curve (ROC) and Area Under the Curve (AUC) with respect to the accuracy of the SenseToKnow app for autism versus non-autism classification | Will be calculated based on data from Baseline/Timepoint 1
  ROC is a graphical plot that illustrates the diagnostic ability of a binary classifier system as its discrimination threshold is varied. AUC measures the area underneath the entire ROC curve.
Sensitivity of SenseToKnow + Parent Survey for autism detection | Will be calculated based on data from Baseline/Timepoint 1
  Sensitivity = #participants positive for autism on both SenseToKnow+Parent Survey and expert clinical diagnosis / # participants positive for autism on both SenseToKnow+Parent Survey and expert clinical diagnosis + #participants negative for autism on SenseToKnow+Parent Survey who were positive for autism by expert clinical diagnosis
Specificity of SenseToKnow + Parent Survey Survey for autism detection | Will be calculated based on data from Baseline/Timepoint 1
  Specificity = #participants negative for autism on both SenseToKnow+Parent Survey and expert clinical diagnosis / #participants negative for autism on both SenseToKnow+Parent Survey and expert clinical diagnosis + #participants positive for autism on SenseToKnow+Parent Survey who were negative for autism by expert clinical diagnosis
Positive Predictive Value of SenseToKnow + Parent Survey (with and without adjustment for population prevalence) | Will be calculated based on data from Baseline/Timepoint 1
  The likelihood that a participant with a positive test result has a diagnosis of autism.
Negative Predictive Value of SenseToKnow + Parent Survey (with and without adjustment for population prevalence) | Will be calculated based on data from Baseline/Timepoint 1
  The likelihood that a participant with a negative test result does not have a diagnosis of autism
Receiver Operating Characteristic Curve (ROC) and Area Under the Curve (AUC) with respect to the accuracy of the SenseToKnow app + Parent Survey for autism versus non-autism classification | Will be calculated based on data from Baseline/Timepoint 1
  ROC is a graphical plot that illustrates the diagnostic ability of a binary classifier system as its discrimination threshold is varied. AUC measures the area underneath the entire ROC curve.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Dawson, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual-level data that meets PHI and IRB confidentiality requirements will be submitted to the NIH/NIMH Data Repository by the end of the grant period.
Supporting Information: Analytic Code
Time Frame: We will submit an electronic version of the final, peer-reviewed work, including the statistical analysis code, to the National Library of Medicine PubMed Central, to be made publicly available no later than 12 months after the official date of publication.
Access Criteria: Publically available via PubMed Central
URL: https://pubmed.ncbi.nlm.nih.gov/